CLINICAL TRIAL: NCT00727623
Title: Prospective Observational Study to Assess Predictors of in Hospital Mortality in STEMI Patients Admitted in Belgian Hospitals
Brief Title: Mortality Analysis of ST Elevation Myocardial Infarction (STEMI) Patients in Belgium
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Belgian Government (Other Government)
Responsible Party: Principal Investigator, M Claeys, Prof dr, Universiteit Antwerpen
Other Study IDs: BIWAC-01
Record Dates: First submitted 2008-07-29; First posted 2008-08-04 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Acute Myocardial Infarction
Keywords: acute coronary syndrome; myocardial infarction; predictors of mortality; reperfusion therapy
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to assess predictors of in-hospital mortality in patients with acute myocardial infarction admitted to Belgian hospitals.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of acute myocardial infarction with ST elevation or left bundle branch blok pattern on ECG

Exclusion Criteria:

* acute myocardial infarction as an acute complication of coronary intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute ST elevation myocardial infarction admitted in Belgian hospitals.
Sampling Method: Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2025-06 (Actual)

PRIMARY OUTCOMES:
all cause mortality | one month

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Claeys, MD.PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Centre Hospitalier de Jolimont, La Louvière, Hainaut, Belgium

REFERENCES:
- [Derived] Gevaert SA, De Bacquer D, Evrard P, Convens C, Dubois P, Boland J, Renard M, Beauloye C, Coussement P, De Raedt H, de Meester A, Vandecasteele E, Vranckx P, Sinnaeve PR, Claeys MJ. Gender, TIMI risk score and in-hospital mortality in STEMI patients undergoing primary PCI: results from the Belgian STEMI registry. EuroIntervention. 2014 Jan 22;9(9):1095-101. doi: 10.4244/EIJV9I9A184. PMID 24457280